## Effects Of Sensory Training and Electrical Stimulation on

## Sole of The Foot Sensations in Patients With Acute Hemiplegia

PT. CANSU HAYIROĞLU YEDITEPE UNIVERSITY 17.02.2020

## Statistical Analysis Plan

In our study; data analysis "Statistical Package for Social Sciences" (SPSS) Version 25.0 program was used. Descriptive statistics, mean  $\pm$  standard deviation (X  $\pm$  SD) or percentages (%), were gathered. The level of significance was accepted as p $\leq$ 0,05. Statistical analysis was performed before and after treatment for parametric and nonparametric data with respectively Paired Sample T-test and Wilcoxon test. An independentsamples t test was used to compare physical features. A Chi-square test was used to assess categorical variables. An independentsamples t test and mann-whitney u test were used to compare of parametric and nonparametric variables between participants before interventions. A Wilcoxon test for non parametric variables and paired-samples t test for parametric variables were used to examine group differences in regard to pre and post test mean scores. A Mc Nemar Test was used to compare before and after treatment for categorical data.